CLINICAL TRIAL: NCT01762930
Title: Study of Field Application of Oral Cholera Vaccine, Shanchol for Use in Developing Country Settings
Brief Title: Field Application of Shanchol in Adults in Bangladesh
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-12030
Record Dates: First submitted 2012-10-16; First posted 2013-01-08 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Other Specified Effects of Reduced Temperature
MeSH Terms: interventions — shanchol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Shanchol stored at 2-8oC (Active Comparator): Vaccines will be stored at 2-8oC before administration.
  Interventions: Drug: Shanchol
- Shanchol stored at 25oC (Experimental): Vaccines will be stored at 25oC for 14 days before administration.
  Interventions: Drug: Shanchol
- Shanchol stored at 37oC (Experimental): Vaccines will be stored at 37oC for 14 days before administration.
  Interventions: Drug: Shanchol
- Shanchol stored at 42oC (Experimental): Vaccines will be stored at 42oC for 14 days before administration.
  Interventions: Drug: Shanchol

INTERVENTIONS:
Drug: Shanchol — Each dose of the vaccine contains inactivated whole cell, heat killed and formalin killed bacteria measured as ELISA Units (EU) of lipopolysaccharide (LPS). It contains formalin-killed V. cholerae Inaba, El Tor biotype (strain Phil 6973; 600 EU); heat-killed V. cholerae Ogawa classical biotype (Cairo 50; 300 EU); formalin killed V. cholerae Ogawa classical biotype (Cairo 50; 300 EU); LPS of heat-killed V. cholerae Inaba, classical biotype (Cairo 48; 300 EU); and formalin killed V. cholerae O139 (4260B; 600 EU).

SUMMARY:
Background:

Cholera is a public health problem globally and in Bangladesh and its prevention is important. Despite recent availability of an effective and affordable oral cholera vaccine (OCV), its field application remains a challenge and needs to be addressed in carefully conducted research studies.There is lack of information on temperature sensitivity and resulting immunogenicity of Shanchol OCV and it is not known if administration of two doses of OCVs, one month apart, instead of currently recommended 14 days, to improve success of vaccination programme will be effective;also if one dose of the vaccine, instead of currently recommended two doses, would result in adequate immune response in population exposed to V. cholerae in an endemic country like Bangladesh.

Objectives:

To determine immunogenicity of Shanchol in adults. when:

1. the vaccine is stored at three defined temperatures(25 oC ,37 oC and 42oC) for 14 days, before putting back in cold box for administration in the field and compare them with the response when the vaccine is stored under currently recommended temperatures.
2. two doses of the vaccine administered one month apart and compared vaccines administered at currently recommended interval of 14 days.
3. a single dose is administered and compare them with responses after recommended two doses.

Methods: The study will be conducted among adults living in the Mirpur community in urban Dhaka, the capital of Bangladesh.Studying safety and acute and long-term immune responses over a period of one year.

Outcome measures/variables:

1. Objective 1: safety and immunogenicity of vaccine in adults after its storage at three defined temperatures (25oC ,37oC and 42oC) by measuring vibriocidal antibody responses and compare them with the findings when the vaccine is stored at currently recommended temperature of 2-8oC (recommended by manufacturer, Shantha Biotechnic).
2. Objective 2: compare vibriocidal responses following administration of two doses of the vaccine one month apart and compare them with vaccination 14 days apart over a period of one year, with study of the memory responses over a one year period as a secondary outcome.
3. Objective 3: compare acute immune responses (vibriocidal antibody) following one and two doses of vaccine, and compare memory response as a secondary outcome measure, over a one year period.

The above information is needed urgently for developing effective vaccination strategies for prevention and control of cholera in endemic countries.

DETAILED DESCRIPTION:
Cholera remains a major cause of morbidity and mortality in Bangladesh and many other endemic countries in the world.The WHO recommends using the cholera vaccine in both epidemic and endemic areas to control outbreaks.An affordable oral vaccine is now available for use in endemic settings; however, successful vaccination remains challenging and expensive due to the need for temperature-controlled distribution systems, which is difficult in most developing countries.Therefore, it would be important to test heat stability of the current vaccines without significantly compromising its safety and efficacy.

In cholera endemic populations their baseline immune responses and memory to the pathogen already exists. Therfore, a single dose of cholera vaccine could act as booster dose eliminating the need for the second dose, saving costs but more importantly significantly improving its delivery to large number of people within a very short time. However, that needs study in endemic countries, such as Bangladesh, to examine both acute and memory responses following a single dose and to determine how long they persist.

In the developing countries such as in Bangladesh, vaccination with two doses can be problematic, with logistic and cost issues. It is also difficult to administer two doses of the vaccine after an interval of 14 days - increasing the interval to one month would be more practical and that would improve coverage of large number of populations. It would, therefore, be important to examine if immunogenicity could be increased when the second dose is administered 30 days following the first dose.

Adult males and females living in the Mirpur community in urban Dhaka will be recruited in the study.The community will be informed by the field staff and interested persons will be recruited according to the inclusion/exclusion criteria.

Eligible participants will receive Shanchol vaccine according to study design. The vaccine comes in single-dose vials and is 1.5 mL in volume.

Group 1: Immunogenicity studies on temperature stability of Shanchol The vaccines will be stored at different temperatures

1a. 25°C for 14 days

1b. 37°C for 14 days and

1c. 42°C for 14 days.

After that vaccine will be stored at the recommended tempature in cold chain until their administration to the participants. The second dose will be administered 14 days after the first dose, as currently recommended. These three groups will be compared to those receiving the same vaccine maintained at standard conditions of 2-8oC.We will enroll 145 participants in each of the four groups (three interventions and a control) i.e. a total of 580 eligible participants. We will measure acute responses to the vaccine by measuring vibriocidal antibodies up to a period of 28 days.

Group 2a: Immunogenicity of two doses of Shanchol given 14 days apart and immunogenicity measured over a one year period Two doses of vaccines, maintained at standard storage condition (2-8oC), will be administered 14 days apart to evaluate the acute and long term immune responses.A total of 145 eligible participants will be studied in this group. We will compare acute and long term immune response among participants in this group with those in Group 2b and Group 3.

Group 2b: Immunogenicity of two doses of Shanchol given 30 days apart and immunogenicity measured over a one year period Two doses of vaccines, maintained at standard storage condition (2-8oC), will be administered 30 days apart to evaluate the acute and long term immune responses. A total of 145 eligible participants will be studied in this group. We will compare acute and long term immune responses in this group with those in Group 2a and Group 3.

Group 3: Immunogenicity of a single dose of Shanchol over a one year period A single dose of the vaccine, maintained at standard temperature (2-8oC), will be administered. The acute and long term immune response would be measured for a one-year period. A total of 145 participants will be enrolled in this group. We will compare immune response among particiupants in this group with those in Groups 2a and 2b.

Duration of the study period for individual participants

The participants in Group 1 will be followed upto 28 days, and remaining groups will be followed up to 1 year.

Surveillance for adverse effects:

The study participants will be monitored after the intervention to assess the safety of the study agent. After each dose of vaccine, the recipients will be followed up for 30 minutes in the clinic and then sent home if they do not have problem. Under the supervision of a clinic physician, trained Research Assistants will visit the participants in their respective homes for the next 3 cosecutive days to record adverse events such as diarrhea, vomiting, nausea and other local and systemic reactions constituting active surveillance. For the next 11 days, passive surveillance will be carried out and participants will be instructed to visit the field clinic if they have any problems. All adverse events during the study period will be recorded and the conditions managed either at the clinic or at the Dhaka Hospital of icddr, b or at other clinics/hospitals depending on the nature and severity of the condition at no costs to the participants. A clinical record form will be used to record all clinical signs and symptoms. For serious adverse events data will be entered onto a separate form.

Study intervention: Oral cholera vaccine, Shanchol Each dose of the vaccine contains inactivated whole cell, heat killed and formalin killed bacteria measured as ELISA Units (EU) of lipopolysaccharide (LPS). It contains formalin-killed V. cholerae Inaba, El Tor biotype (strain Phil 6973; 600 EU); heat-killed V. cholerae Ogawa classical biotype (Cairo 50; 300 EU); formalin killed V. cholerae Ogawa classical biotype (Cairo 50; 300 EU); LPS of heat-killed V. cholerae Inaba, classical biotype (Cairo 48; 300 EU); and formalin killed V. cholerae O139 (4260B; 600 EU).

Storage conditions The vaccine will be stored at 2-8°C under standard conditions (recommended) and in incubators at 25°C, 37 °C and 42°C for 14 days for the study purpose.

Vaccine allocation: The study is an open study although the investigators in the laboratory carrying out the tests will be blinded as the batch of vaccine allocation they are testing. The vaccines will be allocated based on the temperature at which they have been incubated and starting from the lowest 25 oC and then going up finally to 42oC in the different sets of study participants. Each set of vaccines stored at the different temperatures will be given a code (25oC, 37oC and 42oC stored batches).

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy individuals
2. Age: 18-45 years
3. Sex: Both male and female
4. Consent: Written informed consent form for participation in the study

Exclusion Criteria:

1. History of chronic illness, such as TB, hypertension, chronic asthma, diabetes
2. Gastrointestinal disorder such as abdominal pain or cramps, loss of appetite, nausea, vomiting or diarrhoea in the past 7 days
3. Intake of any anti-diarrheal medicine in the past one week or antimicrobial therapy in the past two weeks.
4. Any febrile illness in the past 7 days.
5. Receiving killed oral cholera vaccine any time in the past, and any other live or killed enteric vaccine in the last 4 weeks.
6. Immunocompromising condition or receipt of blood or blood products or parenteral immunoglobulin preparation in the past 3 months.
7. Females of reproductive age who are pregnant at the time of vaccination and follow up (determined by verbal screening e.g last menstrual period (LMP)).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1015 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of Shanchol cholera vaccine | 1 year
  Immunogenicity of Shanchol vaccine will be measured by vibriocidal response in adults storing the vaccine at 2-8 0 c, 25 oC, 37 oC and 42oC

SECONDARY OUTCOMES:
Immunogenicity by vibriocidal response | 1 year
  Vibriocidal responses following administration of two doses of the vaccine will be measured one month apart and 14 days apart with study of memory responses
Acute and memory B and T cell responses | 1 year
  Acute and memory B and T cell responses following administration of one and two doses of Shanchol vaccine will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Amit Saha, M.Med, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal disease Research,Bangladesh, Dhaka, Dhaka Division, Bangladesh

REFERENCES:
- [Result] Kanungo S, Paisley A, Lopez AL, Bhattacharya M, Manna B, Kim DR, Han SH, Attridge S, Carbis R, Rao R, Holmgren J, Clemens JD, Sur D. Immune responses following one and two doses of the reformulated, bivalent, killed, whole-cell, oral cholera vaccine among adults and children in Kolkata, India: a randomized, placebo-controlled trial. Vaccine. 2009 Nov 16;27(49):6887-93. doi: 10.1016/j.vaccine.2009.09.008. Epub 2009 Sep 15. PMID 19761838
- [Result] Alam MM, Riyadh MA, Fatema K, Rahman MA, Akhtar N, Ahmed T, Chowdhury MI, Chowdhury F, Calderwood SB, Harris JB, Ryan ET, Qadri F. Antigen-specific memory B-cell responses in Bangladeshi adults after one- or two-dose oral killed cholera vaccination and comparison with responses in patients with naturally acquired cholera. Clin Vaccine Immunol. 2011 May;18(5):844-50. doi: 10.1128/CVI.00562-10. Epub 2011 Feb 23. PMID 21346055
- [Result] Saha A, Chowdhury MI, Khanam F, Bhuiyan MS, Chowdhury F, Khan AI, Khan IA, Clemens J, Ali M, Cravioto A, Qadri F. Safety and immunogenicity study of a killed bivalent (O1 and O139) whole-cell oral cholera vaccine Shanchol, in Bangladeshi adults and children as young as 1 year of age. Vaccine. 2011 Oct 26;29(46):8285-92. doi: 10.1016/j.vaccine.2011.08.108. Epub 2011 Sep 9. PMID 21907255
- [Derived] Saha A, Khan A, Salma U, Jahan N, Bhuiyan TR, Chowdhury F, Khan AI, Khanam F, Muruganandham S, Reddy Kandukuri S, Singh Dhingra M, Clemens JD, Cravioto A, Qadri F. The oral cholera vaccine Shanchol when stored at elevated temperatures maintains the safety and immunogenicity profile in Bangladeshi participants. Vaccine. 2016 Mar 18;34(13):1551-1558. doi: 10.1016/j.vaccine.2016.02.020. Epub 2016 Feb 16. PMID 26896684